CLINICAL TRIAL: NCT03628703
Title: Using Repetitive Transcranial Magnetic Stimulation to Modulate Response Inhibition in Tourette Syndrome
Brief Title: Response Inhibition in Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIN001 - TAA2018
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Repetitive TMS (Experimental): Repetitive Intermittent Theta-Burst Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive TMS

INTERVENTIONS:
Device: Repetitive TMS — Repetitive Intermittent Theta-Burst Transcranial Magnetic Stimulation over the right Pre-supplementary Motor Area

SUMMARY:
Tics are the hallmark symptoms in Tourette Syndrome. Patients with Tourette Syndrome have difficulties controlling unwanted movements. The ability to control the motor system involves the pre-supplementary motor area (pre-SMA) in the brain. In this study, we will use Transcranial Magnetic Stimulation to modulate the pre-SMA and determine effect on the ability to stop an unwanted action in a behavior task (stop signal task).

ELIGIBILITY:
Inclusion Criteria:

* Tourette Syndrome

Exclusion Criteria:

* Autism spectrum disorder
* Mood disorder
* Epilepsy
* Implanted medical device (e.g. pacemaker, shunt, pumps)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve W. Wu, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repetitive TMS
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Repetitive TMS
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Yale Global Tic Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The score presented is the total tic severity score, ranging from 0 to 50. A score of 0 is when someone has no tics. A score of 50 is the maximal score for someone with multiple severe tics.
  units on a scale | 19.3 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Stop Signal Reaction Time (SSRT)
Description: SSRT measured from modified Slater-Hammel stop signal task performance. The SSRT is calculated by subtracting the average stop signal delay (msec) from the average go-trial reaction time. The SSRT is a measure of inhibitory behavior. The lower the SSRT value means a person is better at inhibitory control. The higher the SSRT value means a person is worse at inhibitory control.
Time Frame: 30 minutes after Repetitive Transcranial Magnetic Stimulation (as it takes about 30 minutes to complete the modified Slater-Hammel stop signal task)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Repetitive TMS
Number analyzed (Participants) | 10
milliseconds
  Before Repetitive TMS | 249 (28.0)
  After Repetitive TMS | 245 (11.2)
Statistical Analysis 1: Comparison: Repetitive TMS; Test type: Superiority; p = 0.49, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Repetitive TMS
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03628703/Prot_SAP_000.pdf